CLINICAL TRIAL: NCT06077565
Title: A General-health-promotion-approach to Promoting Healthier Lives Among Discharged Emergency Department Attendees: A Randomized Clinical Trial
Brief Title: General-health-promotion-approach to Promoting Healthier Lives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GHPED
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Health-risk Behaviours; Non Communicable Diseases
Keywords: general-health-promotion; healthier lives; emergency department
MeSH Terms: conditions — Noncommunicable Diseases; Emergencies | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants will be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications. the research assistant will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so. For the first 6 months of the study period, the research assistant will deliver WhatsApp/WeChat messages about once per week. Follow-up assessment of behavioural changes at 3, 6, and 12 months
  Interventions: Other: foot-in-the-door technique and self-determination theory; Other: Follow-up booster intervention
- Control group (Placebo Comparator): The participants will be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications.The control group participants will receive a brief telephone intervention based on the AWARD model and delivered by the trained research assistant, similar to that delivered to the intervention group. However, the research assistant will simply advise the participants to change their health-risk behaviours and/or adopt a healthy lifestyle practice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: foot-in-the-door technique and self-determination theory — the research assistant will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise or reducing alcohol consumption. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so. Each participant will then receive a brief (approximately 5 minutes), individual intervention with health advice about the selected health-related lifestyle practice. The whole intervention will last approximately 10 minutes, but slightly longer if necessary.
  Arms: Intervention group
Other: Follow-up booster intervention — For the first 6 months of the study period, the research assistant will deliver WhatsApp/WeChat messages about once per week. If a participant does not own a smartphone or is unable to receive WhatsApp/WeChat messages (uncommon in Hong Kong), the research assistant will make a telephone call, instead of sending a message, as a reminder for the participants to adhere to their desirable health-related lifestyle practice. Instant messaging via mobile applications has found to be effective in enhancing treatment compliance.
  Arms: Intervention group
Other: Control group — The control group participants will receive a brief telephone intervention based on the AWARD model and delivered by the trained research assistant, similar to that delivered to the intervention group. However, the research assistant will simply advise the participants to change their health-risk behaviours and/or adopt a healthy lifestyle practice.
  Arms: Control group

SUMMARY:
Aim To examine the effectiveness of a general-health-promotion-approach to help ED attendees change their health-risk behaviours and lead healthier lives.

Hypotheses to be tested The investigators hypothesise that compared with those in the control group, the participants in the intervention group will experience significantly greater success in changing their health-risk behaviours and will have a better health-related quality of life at 6 months follow-up.

DETAILED DESCRIPTION:
Study design A RCT with a two-group pre-test and repeated post-test between- subjects design will be conducted.

Setting:

The setting is the ED of the United Christen Hospital (UCH), one of the major acute care hospitals in Kowloon East cluster in Hong Kong.

Conceptual and theoretical framework:

The proposed intervention is guided by the foot-in-the-door technique, and self-determination theory.

Foot-in-the-door technique The foot-in-the-door technique, which was introduced by Freeman and Fraser, emphasises the notion that individuals who initially comply with a small, easy request are more likely to later comply with a larger request. Compliance with the first request or target increases the individual's confidence and alters their self-perceived capability and willingness regarding further requests or targets. This technique can facilitate the recruitment process and enhance compliance.

Self-determination theory According to self-determination theory, behavioural regulation is more autonomous when it is internalised, as opposed to being regulated by external factors (e.g., orders from family members, friends, or healthcare professionals). Compared with external regulation, autonomous regulation is associated with increased self-efficacy, greater behavioural persistence, longer-term behavioural changes and more positive health behaviour. Autonomy is another influential determinant of behaviour that is emphasised by freedom of choice. There is some evidence that supports a positive association between autonomy and competence, with people who have greater autonomy demonstrating greater competence in achieving behavioural change compared with those with less autonomy. Evidence suggests that patients who have the opportunity to decide on their own treatment may be more eager to comply with instructions. The participants in this proposed study will be allowed to select their priorities in engaging in desirable health-related lifestyle practices after discussion with the research assistant. It is anticipated that the participants will show a greater willingness to adhere to their desired health-related lifestyle practice as a result of this increase in autonomy. Moreover, there is some evidence for a positive association between autonomy and self-efficacy; that is, people who have greater autonomy demonstrate greater self-efficacy for achieving behavioural change. As a result, increased autonomy will facilitate a gradual change in risky behaviours.

Our intervention, therefore, aims to first change the participants' attitudes and their subjective norms through risk communication. By using the foot-in-the-door technique and self-determination theory, it will then enhance the participants' self-efficacy in changing their health-risk behaviours.

Intervention

At the ED All potential participants will be approached by emergency nurses before being discharged home from the ED. The emergency nurse will provide potential participants with a leaflet detailing the nature and purpose of the study. Potential participants can express their willingness to participate in the study by signing an informed consent form. The emergency nurse will then refer the participants to the research assistant. Participants will be informed that they will receive a telephone call from a research assistant within 3 days to evaluate their potential health-risk behaviours and provide them with appropriate health advice to lead healthier lives. The participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications, including (i) 'Move Your Body', (ii) 'Eat Healthy', (iii) 'Live Alcohol Free', and (iv) 'Stay Away from Tobacco', which were developed by the Hong Kong Department of Health.

1. Intervention group Brief intervention via telephone (within 3 days after visiting the ED) The participants will receive a brief intervention using the Ask, Warn, Advise, Refer and Do-it-again (AWARD) model, which was originally developed for primary-care tobacco-cessation interventions. The brief intervention includes the following steps: (1) ask about and assess health-risk behaviours; (2) warn about the high morbidity and mortality risks associated with health-risk behaviours; (3) advise to adopt healthy lifestyle practices to benefit the health of the participant; (4) refer to hotline services on request, such as smoking cessation and alcohol treatment services; and (5) do it again. For the warning message, the research assistant will provide the following standardised message: 'The WHO has identified four major behavioural risk factors, namely, tobacco use, harmful alcohol use, an unhealthy diet and physical inactivity, that contribute substantially to NCDs, which result in high rates of morbidity and mortality.' For the advice step, the research assistant will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise or reducing alcohol consumption. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so. Each participant will then receive a brief (approximately 5 minutes), individual intervention with health advice about the selected health-related lifestyle practice. The whole intervention will last approximately 10 minutes, but slightly longer if necessary. Such a brief intervention will be more feasible for routine use in clinical practice by healthcare professionals after minimal training. Previous clinical trials of smoking cessation have provided strong evidence regarding the effectiveness of brief interventions using the AWARD model.

   At the end of the telephone call, the participants will be informed that throughout the study period, the research assistant will assist in achieving the participant's health-related goals by sending WhatsApp/WeChat messages or via telephone calls.

   Follow-up booster intervention (up to 6 months) For the first 6 months of the study period, the research assistant will deliver WhatsApp/WeChat messages about once per week. If a participant does not own a smartphone or is unable to receive WhatsApp/WeChat messages (uncommon in Hong Kong), the research assistant will make a telephone call, instead of sending a message, as a reminder for the participants to adhere to their desirable health-related lifestyle practice. Instant messaging via mobile applications has found to be effective in enhancing treatment compliance.

   Follow-up assessment of behavioural changes at 3, 6, and 12 months The participants will be assessed to determine their success in changing their targeted health-related lifestyle practice via a phone call at 3, 6, and 12 months.
2. Control group The control group participants will receive a brief telephone intervention based on the AWARD model and delivered by the trained research assistant, similar to that delivered to the intervention group. However, the research assistant will simply advise the participants to change their health-risk behaviours and/or adopt a healthy lifestyle practice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.

Randomisation method To avoid the potential risk of treatment contamination within the ED, randomisation will not be performed there. Instead, the research assistant will input the baseline data collected at the ED directly into the web-based trial entry form linked to a computerised database, and randomisation will then be performed at the Principal Investigator's (PI's) institution by an independent statistician who will have no other involvement in the study. Stratified block randomisation with 1:1 allocation will be conducted using varying block sizes of 2-4 to achieve an appropriate balance of participant numbers between the two groups and to optimise allocation concealment. In addition, the randomization will be stratified by health-risk behaviours (tobacco use, harmful use of alcohol, unhealthy diet, and physical inactivity) to yield a good balance of participant numbers with different lifestyle risk behaviours in the two groups. The subjects will not be able to change group after randomisation.

Sample size G*Power is used to estimate the sample size based on the results of our pilot study. The pilot study showed an approximately 10% between-group difference in reports of successfully abstinence from at least one health-risk behaviour between groups at 12 months. To detect a significant difference in the proportion of participants quitting health-risk behaviours or adopting healthy lifestyle practices between the intervention and control groups, with a power of 80% and a significance level of 5% (2-tailed), at least 199 participants will be needed per group. To account for a potential attrition rate of 30% at the 12-month follow-up assessment, totally 572 participants will be recruited.

According to the Hospital Authority Annual Report,9 there were 140,273 visits in ED of UCH between 2021 and 2022. Furthermore, according to our previous pilot study conducted in ED of UCH, the investigators are confident that they will be able to recruit the required number of participants (N =572) within 15 months.

Data Analysis The baseline characteristics of the two groups will first be compared using the chi-square test for categorical variables and analysis of variance for continuous variables. An intention-to-treat analysis will be used by imputing all non-responses at follow-up by baseline values (i.e. assuming failure or no change after the intervention), to yield more conservative effect size estimates.

SPSS for Windows (SPSS version 26.0; IBM Corp., Armonk, NY, USA) will be used for the quantitative data analysis. Descriptive statistics will be used to calculate the mean, standard deviation, and frequency of the demographic and health-risk behaviour data. The primary analysis including the main effect, i.e., behavioural changes at 6 months in the intervention group versus those in the control group, will be performed using a chi-square test or Fisher's exact test. The secondary analyses will (1) assess the main effect adjusted for baseline differences, (2) assess the secondary outcomes (behavioural changes at 12 months and health-related quality of life at 6 and 12 months), and (3) construct a generalised estimating equation model (GEE). The GEE model will be used to calculate the adjusted odds ratios for the self-reported number of successful health-risk behaviours quit and the number of healthy lifestyles practices engaged in, after adjusting for the baseline demographic and clinical characteristics that show significant differences, and the within-subjects effect of the repeated-measure outcomes (6 and 12 months).

The investigators will conduct a cost-effectiveness analysis CEA using standard methods. The CEA will be populated using empirical 12-month RCT data. An ingredients approach will be used to estimate the cost of the intervention programme, including that of the intervention material (e.g., leaflets and videos), the administration cost, and the time taken to deliver the intervention. The health effectiveness outcomes will include the number of participants who have quit health-risk behaviours at 6 and 12 months and their QALYs.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 18 - 65 years old
* (2) triage as semi-urgent (level 4) or non-urgent (level 5) and will be discharged home after seeking medical attention
* (3) the presence of at least one health risk behaviour (tobacco use, harmful use of alcohol, unhealthy diet and physical inactivity)
* (4) able to communicate in Chinese

Exclusion Criteria:

* (1) poor cognitive state or mental illness
* (2) diagnosed with NCDs and have regular follow-up in outpatient clinics
* (3) participation in another related study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Abstinence from at least 1 health-risk behaviour at 6 months | 6 months
  Abstinence from at least 1 health-risk behaviour between baseline and 6-month follow-up assessed by using a behavioural health-risk factor survey.

SECONDARY OUTCOMES:
Abstinence from at least 1 health-risk behaviour at 12 month | 12 months
  Abstinence from at least 1 health-risk behaviour between baseline and 12-month follow-up assessed by using a behavioural health-risk factor survey.
improved health-related quality of life at 6 months | 6 months
  Participants' the change of health-related quality of life between baseline and 6-month follow-ups will use EuroQol 5-level scale (EQ-5D-5L) to measure the quality of life. It consists of two part. The first part has 5 questions and each question has choices 1 to 5. Large number means a worse outcome in the first part. The second part has one question which is a scale of 0 to 100. Large number means a better outcome in the second part.
improved health-related quality of life at 12 months | 12 months
  Participants' the change of health-related quality of life between baseline and 12-month follow-ups will use EuroQol 5-level scale (EQ-5D-5L) to measure the quality of life. It consists of two part. The first part has 5 questions and each question has choices 1 to 5. Large number means a worse outcome in the first part. The second part has one question which is a scale of 0 to 100. Large number means a better outcome in the second part.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project has been completed and the results of the project has been published
Access Criteria: Request could be sent to Principal Investigator (williamli@cuhk.edu.hk)